CLINICAL TRIAL: NCT05412602
Title: Impact of a Corrective Model of Chiropractic Care on Immune Cell Phenotype and Function
Brief Title: Chiropractic T Cell Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H21-00643
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Intervention; Waitlist Control

STUDY DESIGN:
Intervention Model Description: parallel-arm randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): experimental group will receive 36 chiropractic treatments designed to correct vertebral subluxation over ~12 weeks
  Interventions: Procedure: full spine corrective protocol
- waitlist control (No Intervention): waitlist control will receive no chiropractic interventions and will be reminded that to successfully complete their condition, they do not seek alternative chiropractic treatments

INTERVENTIONS:
Procedure: full spine corrective protocol — 36 chiropractic adjustments over 12 weeks (3 visits per week) with in office spinal traction on the 3D Denneroll Traction Table, as well as supplemental home exercises
  Arms: Intervention

SUMMARY:
Some studies suggest that specific chiropractic care (techniques known as "spinal manipulation therapy") can have benefits to the immune system but studies are scarce, sample sizes small, and methodology and analyses often not of the highest scientific standards. The investigators will example how 36 sessions of chiropractic care over 9-12 weeks can impact immune cell function using a randomized clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18-70.
* Must exhibit vertebral subluxation as measured by a misalignment between one or more vertebrae in relation to normal spinal alignment.
* Have not been sick for the past 3 weeks (immune function).
* Non-smoker.
* Must be able to fast for 10-12 hours.

Exclusion Criteria:

* To have had a chiropractic intervention within the past 6 months.
* To have a condition that may limit the ability to apply a high velocity, low amplitude (HVLA) thrust to the spine such as but not limited to ligament damage, reduced bone density, or other factors that weaken the body's ability to withstand reasonable care (bone cancer, fractures, osteoporosis, etc.)
* To have excessive scoliotic curvature of the spine (> 30º) as measured by identifying the first vertebrae, and the most laterally displaced vertebrae that exhibits tilt below it.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in CD25+ Regulatory T Cell | 12 weeks
  CD25+ Regulatory T Cell count will be measured by surface staining using flow cytometry

SECONDARY OUTCOMES:
Change in CD4+ and CD8+ T cell | 12 weeks
  CD4+ and CD8+ T cell count measured by surface staining using flow cytometry

OTHER OUTCOMES:
Changes in TNF alpha secretion | 12 weeks
  Ex-vivo whole blood culture for either 4 hours in LPS or 24 hours in Poly I:C.
Changes in IFN gamma secretion | 12 weeks
  Ex-vivo whole blood culture for either 4 hours in LPS or 24 hours in Poly I:C.
Change in body mass | 12 weeks
  Body mass in kilograms will be measured by a scale
Change in Blood Pressure | 12 weeks
  Manual blood pressure (systolic and diastolic) in millimetres mercury assessed in the clinic
Change in vertebral subluxation | 12 weeks
  Absolute rotation angle (ARA) of the cervical spine assessed by X-ray
Quality of Life Assessment | 12 weeks
  Differences in quality of life as measured via Oswestry
Quality of Life Assessment | 12 weeks
  Differences in quality of life as measured via SF36
Quality of Life Assessment | 12 weeks
  Differences in quality of life as measured via Neck Disability Index.
Change in Posture | 12 weeks
  Posture analysis as measured by JTech Digital Inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No